CLINICAL TRIAL: NCT02285517
Title: Comparing Mesh and Modified Meek Skin Grafting Techniques in Third Degree Burned Patients Referred to Burn Ward of Khatam-al-anbia Hospital, Irtan
Brief Title: Comparing Modified Meek and Mesh Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahraki, Babak N., M.D. (Individual)
Collaborators: Zahedan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ShahrakiB
Record Dates: First submitted 2014-10-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Third Degree Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified Meek technique (Active Comparator): Intervention: modified Meek skin grafting technique. Patients with third degree of burns without infected wounds are included and the modified Meek results are studied , measured and compared to other group which is operated lesions by mesh technique
  Interventions: Procedure: modified Meek skin grafting technique
- mesh technique (Active Comparator): Intervention: mesh skin grafting technique. patients with third degree of burns without infected wounds are included and the mesh skin grafting technique results are studied , measured and compared to other group which is operated lesions by modified Meek skin grafting technique
  Interventions: Procedure: mesh skin grafting technique

INTERVENTIONS:
Procedure: modified Meek skin grafting technique — patients with third degree of burns and without infected wounds are entered to the study and modified Meek skin grating technique is used to treat them and then the results of the procedure are compared to mesh skin grafting technique results by measuring the square centimeters of healed areas related to the technique
  Arms: modified Meek technique
Procedure: mesh skin grafting technique — patients with third degree of burns and without infected wounds are entered to the study and mesh skin grating technique is used to treat them and then the results of the procedure are compared to modified Meek skin grafting technique results by measuring the square centimeters of healed areas related to the technique
  Arms: mesh technique

SUMMARY:
This is a clinical trial study that compare two plastic surgery techniques in patients with third degree of burning and both techniques are used in all patients but in different areas of burning sites of the patients.

DETAILED DESCRIPTION:
PATIENT REGISTRATION:

The patients are registered after careful examination for third degree of burning and based on the need for skin grafting and of course a written consent were acquired. Excluded patients were those with an infected lesion or those who did not allow us to enter them into the study.

Progression of the treatment results of both techniques were visited by the surgeon regularly.

At the end of the study the data were checked with other similar studies. The acquired data were compared to other external data sources via medical records.

There were two standard operating techniques: modified meek skin grafting technique and mesh skin grafting technique.

The data was analyzed by chi-square and t-test.

ELIGIBILITY:
Inclusion Criteria:

* third degree of burning

Exclusion Criteria:

* infected lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
measuring the size and speed of healing areas under treatment with two different skin graft techniques in a fourteen month period | up to Fourteen months
  Comparing recovering areas operated by two different techniques: square centimeter was the scaling measure

CONTACTS AND LOCATIONS:
Overall Officials: MOSTAFA DAHMARDEHEI, M.D, Principal Investigator — Zahedan University of Medical Sciences; BABAK Na SHAHRAKI, M.D, Principal Investigator — PRIVATE OFFICE

REFERENCES:
- [Background] 6. Hubley P. Review: evidence on dressings for superficial burns is of poor quality. Evid Based Nurs. 2009; 12(3): 78. 7. Jackson D. The diagnosis of the depth of burning. Br J Surg. 1953; 40(164): 558-96. 8. Kreise RW, Mackie DP, Hermans RP and Vlomans AR. Expansion techniques for skin grafts: comparison between mesh and Meek island (sandwich-) grafts. Burns. 1994; 20(1): s39-s42. 9. Jackson D, Topley E, Carson JS. Primary excision and grafting of large burns. Ann Surg. 1960; :152-167. 10. Macmillan BG. Early excision of more than 25% of budy surface in the extensively burned patients. Arch Surg. 1958; 77: 369. 11. Torpy JM, Lynm C, Glass RM. JAMA patient page. Burn injuries. JAMA. 2009; 302(16): 1828. 12. Meek CP. Successfull microdermagrafting using the Meek-wall microdermatome. Am J Surg. 1958; 96(4): 557-558.
- [Background] 13. Lumenta DB, Kamolz LP, Frey M. Adult burn patients with more than 60% TBSA involved-Meek and other techniques to overcome restricted skin harvest availability--the Viennese Concept. J Burn Care Res. 2009; 30(2): 231-42. 14. Raff T, Hartmann B, Wagner H, Germann G. Experience with the modified Meek technique. Acta Chir Plast. 1996; 38(4): 142-146. 15. Kopp J, Magnus Noah E, Rubben A, et al. Radical resection of giant ongenital melanocytic nevus and reconstruction with meek-graft covered integra dermal template. Dermatol Surg. 2003; 29: 653-657. 16. Hsieh CS, Schuong JY, Huang WS, Huang TT. Five years' experience of the modified Meek technique in the management of extensive burns. Burns. 2008; 34(3): 350-354. 17. Wang Zy, He CP, Luo XL, Wang FS. [Clinical application of Meek skin grafting technique] Chinese [Abstract]. Nan Fang Yi Ke Da Xue Xue Bao. 2006; 26(5): 678-9,682.
- [Background] 18. Holmes JH, Honari S. Excision and grafting of the large burn wound. Prob Gen surg. 2003; 20: 47. 19. Menon S, Li Z, Harvey JG and Holland AJ. The use of the Meek technique in conjunction with cultured epithelial autograft in the management of major paediatric burns. Burns. 2013; 39(4): 674-9. 20. Lin C, Chen GX, Zhang P, Lu CJ, Xu JJ, Luo X, Liu ZJ. [Comparison of cost between two ways of skin grafting in the treatment of patients with extensive deep burn] Chinese [Abstract]. Zhonghua Shao Shang Za Zhi. 2009; 25(4): 286-8. 21. Kreis RW, Mackie DP, Hermans RP and Vloemans AR. Expansion techniques for skin grafts: comparison between mesh and Meek island (sandwich-) grafts. Burns. 1994; 20(1): 39-42. 22. Lari AR, Gang RK. Expansion technique for skin grafts (Meek technique) in the treatment of severely burned patients. Burns. 2001; 27(1): 61-66.
- [Result] 1. Endorf FW, Gibran NS. Burns. In: Brunicardi FC, Andersen DK, Billar TR, editors. Schwartz's principles of surgery. 9th ed. New York (USA): McGraw Hill; 2010: 197-206. 2. McGwin G, George RL, Cross JM, et al. Improving the ability to predict mortality among burn patients. Burns. 2008; 34: 320. 3. Ramos CG. Management of fluid and electrolyte disturbances in the burn patient. Annals of Burns and Fire Disasters 2000; 8(4): 21. 4. Wray CJ, Mayes T, Khoury J, Warden GD, Gottschlich M. The 2002 Moyer Award. Metabolic effects of vitamin D on serum calcium, magnesium, and phosphorus in pediatric burn patients.J Burn Care Rehabil. 2002; 23(6): 416-23. 5. Potokar T, Chamania S, Ali S. International network for training, education and research in burns. Indian J Plast Surg 2007;40:107